CLINICAL TRIAL: NCT05550974
Title: Articulating Laparoscopic Instrument Assisted Minimally Invasive Upper GastroIntestinal Surgery: AMUGIS Registry
Brief Title: Articulated Laparoscopic Instruments Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0414
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Gastric Cancer
Keywords: Articulated laparoscopic instruments; gastrointestinal surgery; complication
MeSH Terms: conditions — Stomach Neoplasms | interventions — Minimally Invasive Surgical Procedures; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (6):
- LC: laparoscopic surgery using conventional laparoscopic instruments
  Interventions: Device: Minimally Invasive Surgery
- LW: Using wristed laparoscopic instruments (Artisential Maryland dissector, Artisential Fenestrated gasper)
  Interventions: Device: Minimally Invasive Surgery
- RC: Conventional robotic surgery
- RSS: Use of singlesite system for reduced port robotic surgery
- RSP: Use of da Vinci SP system for reduced port robotic surgery
- RRI: A new surgical robot Revo-i developed by Meerae company in Korea

INTERVENTIONS:
Device: Minimally Invasive Surgery — gynecological, urologic, thoracic, plastic and reconstructive and ENT etc. endoscopic and laparoscopic surgical procedures
  Other Names: Laparoscopic Surgery
  Groups: LC; LW

SUMMARY:
Recently, with the development of minimally invasive surgery and the development of instruments, laparoscopic and robotic surgery are increasing, and laparoscopic and robotic surgery are evolving. The association between the new surgical instruments used in each upper gastrointestinal surgery and the results has been traditionally analyzed through the learning curve, and in addition, the study aims to collect and analyze the utilization of the instrument and surgical results prospectively through surgical video analysis.

DETAILED DESCRIPTION:
Prior to surgery, all patients subject to the study are explained and informed of the prior consent form of prior consent is delivered. During surgery, video recording is performed to check the type of surgical instrument, the time of use, and the event that occurred during surgery. After surgery, the morbidity after surgery will be monitored and recorded. Additional morbidity will be recorded one to three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients with gastric cancer shcedulled for gastrectomy

Exclusion Criteria:

Vulnerable subject (illiterate, pregnant)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer scheduled to undergo gastrectomy in high volume center
Sampling Method: Non-Probability Sample
Enrollment: 1155 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
complication | 1 month after surgery
  One of the most important surgical outcome, complication will be measured at 1 month after surgery

SECONDARY OUTCOMES:
Surgical outcome: operative time(min) | 1 month after surgery
Surgical outcome: bleeding(ml) | 1 month after surgery
  operative time(min), bleeding(ml), pain score, hospital stay(day), readmission rate(%), serum CRP(mg/L), serum Amylase(U/L), serum Lipase(U/L), Drain Amylase(U/L), Drain Lipase(U/L)
Surgical outcome: pain score | 1 month after surgery
  Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Surgical outcome: hospital stay(day) | 1 month after surgery
Surgical outcome: readmission rate(%) | 1 month after surgery
Surgical outcome: serum CRP(mg/L) | 1 month after surgery
Surgical outcome: serum Amylase(U/L) | 1 month after surgery
Surgical outcome: serum Lipase(U/L) | 1 month after surgery
Surgical outcome: Drain Amylase(U/L) | 1 month after surgery
Surgical outcome: Drain Lipase(U/L) | 1 month after surgery
Duration of use for each surgical instruments | during the operation
  Duration for each surgical instruments
number of use for each surgical instruments | during the operation
  number of use for each surgical instruments

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Il Kim, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No